CLINICAL TRIAL: NCT06485089
Title: Effects of Tirzepatide on Blood, Imaging and Breast Tissue Biomarkers in Women With Obesity and Other Risk Factors for Breast Cancer
Brief Title: Effects of Tirzepatide on Blood, Imaging and Breast Tissue Biomarkers
Status: Active, not recruiting | Type: Observational
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Carol Fabian, MD, Professor, University of Kansas Medical Center
Other Study IDs: STUDY00160627
Record Dates: First submitted 2024-06-20; First posted 2024-07-03 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Obesity; Breast Cancer Risk
MeSH Terms: conditions — Obesity | interventions — Tirzepatide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, stool, benign breast tissue
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- women using tirzepatide for weight loss: Women attending the University of Kansas Medical Center (KUMC) Weight Management Clinic
  Interventions: Drug: tirzepatide

INTERVENTIONS:
Drug: tirzepatide — Women taking tirzepatide as part of standard care in the Weight Managment Clinic

SUMMARY:
Evaluation of biomarkers for risk of developing breast cancer in women with obesity who are using tirzepatide to achieve weight loss.

DETAILED DESCRIPTION:
Women who are scheduled to take tirzepatide for weight loss will be assessed before and after taking drug for change in risk biomarkers. These include mammography, DXA scan, blood draw, and random periareolar fine needle aspiration (RPFNA) for acquisition of benign breast tissue.

ELIGIBILITY:
Inclusion Criteria:

* • BMI 30-45 kg/m2

  * Female
  * Insurance approved or likely approved for tirzepatide clinical use *
  * Additional risk factors for breast cancer other than obesity (any one or more) First or second degree with breast cancer Known high density on mammogram (heterogenous or extremely dense) Prior biopsy showing atypical hyperplasia or LCIS Prior treated DCIS Known carrier breast cancer predisposition gene mutation or known mutation in family member .

    2- fold or higher estimated 10 year or lifetime risk compared to population by standard risk model (BCRAT, BCSC, IBIS

Exclusion Criteria:

* • Subglandular breast implants (women with subpectoral implants are eligible if C cup or greater; breast can easily be pulled off the chest wall; and with approval of PI)

  * Clinical contra-indication to incretin mimetics
  * Insurance/third party has denied coverage and participant does not wish to do self-pay.
  * Child-bearing potential and not on contraceptives
  * Prior invasive breast cancer
  * Currently taking any of the following medications: insulin, tamoxifen, raloxifene, letrozole, arimidex, exemestane, incretin mimetics.

Ages: 40 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Must be biologically female
Study Population: Women attending the KUMC Weight Management Clinic and approved or likely to be approved to start a clinical standard of care regimen of tirzepatide for weight loss.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-09-14 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Feasibility of design as assessed by accrual rate of 1 or more per month over 12 months | 12 months
  Accrual defined as signed consent and ompleting baseline proceedures
Completion rate of 70% or more | 6 months
  Completion of procedures for biomarker assessment after 3-6 months of tirzeptide

SECONDARY OUTCOMES:
Change in mammographic fibroglandular volume | 6 months
  as measured by Volpara software baseline and 6 months
Change in benign breast tissue proliferation | 3-6 months
  Difference in baseline and off study Ki-67 in women with baseline Ki-67 of 1 % or higher
Change in benign breast tissue estrogen response and ELF5 gene expression | 3-6 months
  Difference in baseline and off study mRNA
Assessment of GIP-R expression in breast tissue | 3-6 months
  GIP- R mRNA and protein
Change in selected adipokines, cytokines, hormones, IGF-1, alpha klotho | 3-6 months
  change in blood levels with assays primarily by ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Carol J Fabian, MD, Principal Investigator — University of Kansas Medical Center
Locations (2):
- United States (2):
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kansas Medical Center Breast Cancer Prevention Center, Westwood, Kansas

IPD SHARING:
Plan to Share IPD: No
Limited number of participants increases risk of identification of individuals